CLINICAL TRIAL: NCT01401764
Title: Randomized, Double Blind, Crossover, Single Centre Study Comparing The Tolerability Of Three Excipient Formulations Administered Subcutaneously To Healthy Subjects
Brief Title: Study Comparing The Tolerability Of Three Excipient Formulations Administered Subcutaneously To Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: B2271022; 2011-000419-15
Record Dates: First submitted 2011-07-12; First posted 2011-07-25 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platform II, PASS, ARG 100 (Other)
  Interventions: Other: Formulation buffers

INTERVENTIONS:
Other: Formulation buffers — Platform II: Histidine, Polysorbate-80 PASS: Phosphate, Arginine, NaCl ARG 100: Phosphate, 100 mM Arginine

SUMMARY:
The purpose of the study is to compare local pain experienced after subcutaneous injection of three excipient buffers for delivering protein drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects(no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory.
* Body mass index of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Acute disease state (e.g., nausea, vomiting, fever, or diarrhea) within 7 days before study day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Relative perception of pain of platform II versus PASS using a likert scale | 0 minute after injections
Relative perception of pain of platform II versus PASS using a likert scale | 2 minute after injections
Relative perception of pain of PASS versus Arg 100 using a likert scale | 0 minute after injections
Relative perception of pain of PASS versus Arg 100 using a likert scale | 2 minute after injections
Perception of pain of Platform II, PASS and Arg 100 using VAS scale. | 0 minute after injections
Perception of pain of Platform II, PASS and Arg 100 using VAS scale. | 2 minute after injections
Perception of burning of Platform II, PASS and Arg 100 using VAS scale. | 0 minute after injections
Perception of burning of Platform II, PASS and Arg 100 using VAS scale. | 2 minute after injections

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, Study Director — Ablynx, a Sanofi company
Locations (1):
- Investigational Site, Brussels, Belgium